CLINICAL TRIAL: NCT04930315
Title: SHR-1210 Combined With Apatinib Mesylate in the Perioperative Therapy for Technically Resectable Hepatocellular Carcinoma
Brief Title: SHR-1210 Combined With Apatinib Mesylate in the Perioperative Therapy for Hepatocellular Carcinoma
Acronym: CAPT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-11
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; neoadjuvant therapy; adjuvant therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- neoadjuvant and adjuvant group (Experimental): Preoperative：Camrelizumab ：200mg, iv, d1, q2w, 4 cycles；apatinib：250mg, po, qd, q2w, 3 cycles Operation Postoperation 4-8 weeks，Camrelizumab ：200mg, iv, d1, q2w, Up to 8 cycles
  Interventions: Drug: Apatinib Mesylate; Drug: Camrelizumab
- adjuvant group (Active Comparator): Operation Postoperation 4-8 weeks，Camrelizumab ：200mg, iv, d1, q2w, Up to 12 cycles
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Apatinib Mesylate — 250mg, po, qd, q2w in neoadjuvant and adjuvant group, before surgery
  Arms: neoadjuvant and adjuvant group
Drug: Camrelizumab — 200mg, iv, d1, q2w, both in two groups

SUMMARY:
The purpose of this study was to compare the efficacy and safety of camrelizumab + apatinib mesylate neoadjuvant therapy combined with camrelizumab adjuvant therapy and camrelizumab adjuvant therapy alone in patients with technically resectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
The purpose of this study was to compare the efficacy and safety of camrelizumab + apatinib mesylate neoadjuvant therapy combined with camrelizumab adjuvant therapy and camrelizumab adjuvant therapy alone in patients with technically resectable hepatocellular carcinoma. There are two groups:

1. Neoadjuvant and adjuvant group: (1) Preoperative：Camrelizumab ：200mg, iv, d1, q2w, 4 cycles；apatinib：250mg, po, qd, q2w, 3 cycles; (2) Operation; (3) Postoperation 4-8 weeks，Camrelizumab ：200mg, iv, d1, q2w, Up to 8 cycles.
2. Adjuvant group: (1) Operation; (2) Postoperation 4-8 weeks，Camrelizumab ：200mg, iv, d1, q2w, Up to 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* 1)Aged 18-70 years old, both genders.
* 2)Histologically confirmed diagnosis of HCC or strictly consistent with the clinical diagnostic criteria for HCC according to AASLD guideline
* 3)BCLC stage was B / C, or CNLC stage was IIa-IIIb, but technically resectable (the number of tumors was less than 7, accompanied by ipsilateral portal vein or hepatic vein tumor thrombus formation, but no main portal vein, contralateral portal vein, contralateral hepatic vein or inferior vena cava tumor thrombus, no extrahepatic metastasis, estimated residual liver volume > 30% [if patients with liver fibrosis, residual liver volume > 40%])
* 4)At least one measurable lesion that meet the mRECIST standard, and the lesion has not received radiotherapy, or local treatments
* 5)Child-Pugh score: A grade
* 6)ECOG PS 0-1 points.
* 7)The function of vital organs meets the following requirements (excluding the use of any blood component and cell growth factor within 14 days) :

  1. Neutrophils ≥1.5×109/L
  2. Platelet count ≥100×109/L
  3. Hemoglobin ≥90g/L
  4. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN)
  5. AST or ALT levels ≤ 1.5 times the upper limit of normal value (ULN);
  6. Serum albumin ≥ 30 g / L
  7. Thyroid stimulating hormone (TSH) ≤ ULN
  8. Subjects who did not receive anticoagulant therapy: International standardized ratio INR or Partial thromboplastin time APTT≤1.5×ULN; subjects received prophylactic anticoagulant therapy, INR≤1.5×ULN and APTT ≤ ULN within 14 days before the start of study treatment;
  9. Serum creatinine (SCr) ≤ 1.5 times upper limit of normal value (ULN) and creatinine clearance ≥60 ml/min (Cockcroft-Gault formula)
* 8)If HBsAg (+) and / or anti HCV (+), according to the results of HBV DNA or HCV RNA detection, antiviral therapy should be carried out according to the standard
* 9)Women of childbearing age should with negative serum or urine pregnancy tests within 14 days prior to study inclusion and who must be non-lactating, and patient should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during and within 60 days of the end of medication
* 10)Males with partner of childbearing age should agree to use contraceptives during the study period and for 120 days after the end of the study period;
* 11)Subjects have good compliance and cooperate with the follow-up.

Exclusion Criteria:

* 1)Known hepatobiliary cell carcinoma, mixed cell carcinoma and fibre-lamellar cell carcinoma;
* 2)Co-infection with hepatitis B and C, or co-infection with hepatitis B and D
* 3)Active malignancies other than HCC within 5 years or concurrently, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix and papillary thyroid cancer
* 4)Subjects has received radical hepatectomy, systemic anticancer therapy for HCC (mainly including systemic chemotherapy, molecular targeted therapy and CTLA-4, PD-1 / PD-L1 monoclonal antibody immunotherapy) and local treatment for liver, including TACE, TAE, tare or local ablation, radiotherapy, etc
* 5)Presence of the following within 3 months prior to study entry: myocardial infarction, severe unstable angina, NYHA class 2 or higher cardiac insufficiency, poorly controlled arrhythmias, symptomatic congestive heart failure, cerebrovascular accident.
* 6)Having hypertension that cannot be well controlled by antihypertensive drug therapy (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);Previous history of hypertension crisis or hypertensive encephalopathy;
* 7)Active pulmonary tuberculosis or pulmonary tuberculosis history
* 8)Subject has any active autoimmune disease or history of autoimmune disease (such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or childhood asthma have been completely relieved and may be included as adults without any intervention;Asthma requiring medical intervention with bronchodilators will not be included);
* 9)Interstitial lung disease history or non-infectious pneumonia requiring oral or intravenous steroid therapy
* 10)Subjects are receiving immunosuppressive, or systemic, or absorbable local hormone therapy for immunosuppression purposes (>10mg/ day prednisone or other therapeutic hormones) and continue to receive such therapy within 2 weeks prior to enrollment;
* 11)Abnormal coagulation (INR > 1.5 or APTT > 1.5 x ULN) with bleeding tendency or on thrombolytic or anticoagulant therapy
* 12)The presence of clinically significant bleeding symptoms or a definite bleeding tendency within 3 months prior to study entry, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood +++ or more at baseline, or vasculitis. Gastroscopy was performed if fecal occult blood was positive at baseline, or if it was an observable bloody stool. If gastroscopy indicated severe esophageal varices, it could not be included
* 13)Known hypersensitivity to apatinib, camrelizumab or drug excipients; or severe allergic reactions to other monoclonal antibodies
* 14)Subject has active infection or unexplained fever of >38.5 degrees during screening and before first administration (subject's fever due to tumor can be enrolled according to the investigator's judgment);
* 15)Grade III or above myelosuppression (WBC < 1.9) × 109 / L, hemoglobin lower than 79 g / L, platelet lower than 49 g / L × 109/L）
* 16)Severe liver dysfunction, serum albumin less than 28 g/L, or serum bilirubin more than 50 μmol/L, or serum alanine transferase was 1.5 times higher than normal
* 17)HIV positive (HIV 1/2 anti-body)
* 18)Live vaccine is administered less than 30 days before or possibly during the study period;
* 19)The subject has a known history of psychotropic substance abuse, alcohol abuse or drug abuse;
* 20)Researchers think that should be left out in this study, the researchers determine, for example, the subjects have other factors that may result in this study were forced to midway termination, such as, other serious disease (including mental illness) need to merge treatment, there are serious abnormal laboratory examination, accompanied by factors such as family or society, will affect the safety of the subjects, or information and the collection of the sample.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
1-year tumor recurrence-free rate | Up to one years
  The proportion of patients who had tumor recurrence (local, regional or distant) or death within 1 year after surgery, whichever occurred first

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years.
  Overall survival (OS) refers to the time from enrollment to death due to any cause.
Recurrence free survival (RFS) | Up to 1 years
  From radical resection to the date of the first documented tumor into recurrence or death from any cause, whichever occurred first
1-year survival rate | Up to 1 years
  The proportion of patients without death within 1 year after randomization
R0 resection rate | Up to 2 years.
  The proportion of patients with negative resection margin among patients undergoing surgery
Major pathological response (MPR) | Up to 2 years.
  Number of participants experiencing the percentage of the non-viable cancer cells (necrotized or fibrotized) out of the surface expression of the total tumor area is <10%
Pathological Complete Response (pCR) | Up to 2 years.
  After neoadjuvant therapy, no evidence of malignant histology was found in the pathological examination of primary tumor or only carcinoma in situ was found
Surgical resection rate | Up to 2 years.
  the proportion of patients who can accept surgical resection after neoadjuvant therapy
Adverse events | Safety evaluation was done continuously during treatment by using CTCAE 5.0
  Time Frame: 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Dr., Principal Investigator — Zhejiang University; Xueli Bai, Dr., Principal Investigator — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No